CLINICAL TRIAL: NCT04454229
Title: The Use of Penicillin Allergy Clinical Decision Rule to Enable Direct Oral Penicillin Challenge - An International Multicenter Randomized Control Trial - The PALACE Study
Brief Title: The Use of Penicillin Allergy Clinical Decision Rule to Enable Direct Oral Penicillin Challenge
Acronym: PALACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Austin Health (Other Government)
Responsible Party: Principal Investigator, Ana Copaescu, Physician-Scientist Immunology and Allergy, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PALACE1
Record Dates: First submitted 2020-06-25; First posted 2020-07-01 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Hypersensitivity, Immediate; Hypersensitivity, Delayed; Hypersensitivity Response
Keywords: penicillin; Low Risk allergy; direct oral challenge; standard of care; outpatient clinic
MeSH Terms: conditions — Hypersensitivity, Immediate; Hypersensitivity, Delayed | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Direct oral challenge in patients with PEN-Fast less than 3
  Eligible patients referred to the outpatient clinic reporting a penicillin allergy will be identified and assessed with a standard clinical history and the calculation of the PEN-FAST score. PEN-FAST is a three-point clinical assessment tool recently externally validated in a multicenter study, with a PEN-FAST score of < 3 associated with 96.7% negative predictive value.
  Intervention:
  The patient will receive a single dose of oral penicillin, following baseline vital signs (i.e. temperature, heart rate, blood pressure, respiratory rate, skin check).
  Nursing staff will repeat vital signs as needed and after oral challenge while observing for signs of an immune mediated adverse reaction.
  If at any stage an antibiotic associated adverse event is noted, standard of care treatment is offered by the attending clinicians (ex. adrenalin for immediate hypersensitivity reaction).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Direct oral antibiotic challenge (Experimental): Direct oral antibiotic (penicillin) challenge in patients with PEN-Fast less than 3.
  Interventions: Other: Direct oral penicillin challenge
- Standard of care (Active Comparator): Standard of care: skin testing and, if negative, oral challenge.
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Direct oral penicillin challenge — The patient will receive a single dose of oral penicillin, following baseline vital signs.
  Arms: Direct oral antibiotic challenge
Other: Standard of care — Routine management as per the treating clinicians that include skin prick and intradermal beta-lactam testing, followed by oral penicillin challenge in the setting of negative skin testing.
  Arms: Standard of care

SUMMARY:
Whilst validated tools exist to enable inpatient penicillin assessment and de-labelling, limited evidence is available regarding the safety and efficacy in the outpatient clinic. The ability to deliver point-of-care penicillin allergy testing for a large cohort of patients, without skin testing, will improve patient access to testing and utilization of preferred penicillin antibiotics.

DETAILED DESCRIPTION:
Patient-reported penicillin allergies result in poor health outcomes for patients and drive inappropriate antibiotic prescribing, antimicrobial resistance and healthcare costs. Our group has internally and externally validated a novel penicillin allergy clinician decision rule (PEN-FAST) that is able to identify low risk penicillin allergies with a negative predictive value of 96% (95%; 94-98%). Therefore, whilst validated tools exist to enable inpatient penicillin assessment and de-labelling, limited evidence is available regarding the safety and efficacy in the outpatient clinic. The ability to deliver point-of-care penicillin allergy testing for a large cohort of patients, without skin testing, will improve patient access to testing and utilization of preferred penicillin antibiotics.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients referred to the outpatient allergy clinic for a penicillin allergy history;
2. Willing and able to give consent.

Exclusion Criteria:

1. Patient age is < 18 years;
2. Patients with a PEN-FAST score less than 3
3. Pregnancy;
4. Any other illness that, in the investigator's judgement, will substantially increase the risk associated with subject's participation in this study;
5. Patients with history of type A adverse drug reaction, drug-associated anaphylaxis, idiopathic urticaria/anaphylaxis, mastocytosis, serum sickness, blistering skin eruption or acute interstitial nephritis;
6. Patients where the allergy history was not able to be confirmed with patient;
7. Patients on concurrent antihistamine therapy;
8. Patients receiving more than stress dose steroids (i.e. > 50mg QID hydrocortisone [or steroid equivalent]).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-02 (Actual)

PRIMARY OUTCOMES:
The difference in the proportion of positive oral challenges (i.e. immune-mediated reaction) | up to 48H after oral challenge

SECONDARY OUTCOMES:
Proportion of patients referred to the outpatient allergy clinic that are eligible for intervention (i.e randomization) as per protocol [Eligibility to screened ratio] | Before randomization
Feasibility of recruitment defined as the proportion of patients consenting to participate in the study as per protocol from eligible patients. [Recruitment to eligibility ratio]. | Before randomization
Feasibility of intervention delivery defined as the proportion of patients randomized to the intervention arm who had the intervention delivered as per protocol. [Intervention to recruitment ratio] | Before randomization
The proportion of patients with a penicillin allergy who experience an antibiotic associated immune mediated adverse event OR severe adverse drug reaction as per protocol definitions. | Up to 48h after the drug challenge
The proportion of patients with a penicillin allergy who experience an antibiotic associated non-immune mediated adverse event. | Up to 48h after the drug challenge
The proportion of patients that will respect the protocol (protocol compliance) | Up to 48h after the drug challenge
Proportion of patient with positive Penicillin Skin Testing | Up to 48h after the drug challenge
Proportion of patients with non-immune mediated positive oral provocation | Up to 48h after the drug challenge
Proportion of patients with severe adverse reaction - anaphylaxis/death | Up to 48h after the drug challenge
Time from randomization to delabelling | Up to 48h after the drug challenge
Number of appointments required for Penicillin delabelling | Up to 48h after the drug challenge
Assessment with the Pre-Questionnaire and the 6 months follow-up Questionnaire | Up to 6 months after the drug challenge

CONTACTS AND LOCATIONS:
Locations (6):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Australia (3):
  - Austin Health, Heidelberg, Victoria
  - Peter MacCallum Cancer Center, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
- McGill University Health Centre (MUHC), Montreal, Quebec, Canada

REFERENCES:
- [Result] Trubiano JA, Vogrin S, Chua KYL, Bourke J, Yun J, Douglas A, Stone CA, Yu R, Groenendijk L, Holmes NE, Phillips EJ. Development and Validation of a Penicillin Allergy Clinical Decision Rule. JAMA Intern Med. 2020 May 1;180(5):745-752. doi: 10.1001/jamainternmed.2020.0403. PMID 32176248
- [Result] Devchand M, Urbancic KF, Khumra S, Douglas AP, Smibert O, Cohen E, Sutherland M, Phillips EJ, Trubiano JA. Pathways to improved antibiotic allergy and antimicrobial stewardship practice: The validation of a beta-lactam antibiotic allergy assessment tool. J Allergy Clin Immunol Pract. 2019 Mar;7(3):1063-1065.e5. doi: 10.1016/j.jaip.2018.07.048. Epub 2018 Aug 29. PMID 30172019
- [Result] Trubiano JA, Smibert O, Douglas A, Devchand M, Lambros B, Holmes NE, Chua KY, Phillips EJ, Slavin MA. The Safety and Efficacy of an Oral Penicillin Challenge Program in Cancer Patients: A Multicenter Pilot Study. Open Forum Infect Dis. 2018 Nov 17;5(12):ofy306. doi: 10.1093/ofid/ofy306. eCollection 2018 Dec. PMID 30547046
- [Derived] Copaescu AM, Vogrin S, Douglas A, Turner NA, Phillips EJ, Holmes NE, Trubiano JA. Risk of Self-Reported Penicillin Allergy Despite Removal of Penicillin Allergy Label: Secondary Analysis of the PALACE Randomized Clinical Trial. JAMA Netw Open. 2024 Aug 1;7(8):e2429621. doi: 10.1001/jamanetworkopen.2024.29621. PMID 39145980
- [Derived] Copaescu AM, Vogrin S, James F, Chua KYL, Rose MT, De Luca J, Waldron J, Awad A, Godsell J, Mitri E, Lambros B, Douglas A, Youcef Khoudja R, Isabwe GAC, Genest G, Fein M, Radojicic C, Collier A, Lugar P, Stone C, Ben-Shoshan M, Turner NA, Holmes NE, Phillips EJ, Trubiano JA. Efficacy of a Clinical Decision Rule to Enable Direct Oral Challenge in Patients With Low-Risk Penicillin Allergy: The PALACE Randomized Clinical Trial. JAMA Intern Med. 2023 Sep 1;183(9):944-952. doi: 10.1001/jamainternmed.2023.2986. PMID 37459086
- [Derived] Copaescu AM, James F, Vogrin S, Rose M, Chua K, Holmes NE, Turner NA, Stone C, Phillips E, Trubiano J. Use of a penicillin allergy clinical decision rule to enable direct oral penicillin provocation: an international multicentre randomised control trial in an adult population (PALACE): study protocol. BMJ Open. 2022 Aug 8;12(8):e063784. doi: 10.1136/bmjopen-2022-063784. PMID 35940831

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-12-10): https://cdn.clinicaltrials.gov/large-docs/29/NCT04454229/SAP_002.pdf